CLINICAL TRIAL: NCT00010140
Title: A Multicenter Randomized Trial of Sequential Epirubicin and Docetaxel Versus Epirubicin in Node Positive Postmenopausal Breast Cancer Patients
Brief Title: Epirubicin and Tamoxifen With or Without Docetaxel in Treating Postmenopausal Women With Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Collaborative Cancer Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068450; ICCG-C/14/96; EU-20040
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2005-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen by the tumor cells. Combining chemotherapy with hormone therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of epirubicin and tamoxifen with or without docetaxel in treating postmenopausal women who have breast cancer that has spread to the lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the impact of adjuvant epirubicin with or without docetaxel and concurrent or sequential tamoxifen on time to relapse and overall survival in postmenopausal women with node-positive breast cancer.
* Compare the toxic effects of these regimens in this patient population.
* Compare the quality of life in terms of shift in long term toxicity and differences in recuperation in women treated with these regimens.
* Compare the incidence of thromboembolic events during the first 9 months of study and the influence of such events on compliance in women treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to one of two adjuvant chemotherapy treatment arms within 30 days after surgery.

* Arm I: Patients receive adjuvant epirubicin IV on days 1 and 8. Treatment continues every 28 days for 6 courses.
* Arm II: Patients receive adjuvant epirubicin IV on days 1 and 8. Treatment continues every 28 days for 3 courses. Patients then receive docetaxel IV over 1 hour on day 1. Treatment continues every 21 days for 3 courses.

Patients may be further randomized to one of two tamoxifen arms. Patients not randomized to the tamoxifen arms receive oral tamoxifen daily for 5 years concurrently with adjuvant chemotherapy.

* Arm I: Patients receive tamoxifen as above concurrently with adjuvant chemotherapy.
* Arm II: Patients receive sequential tamoxifen as above after completion of adjuvant chemotherapy.

Quality of life is assessed at baseline, 9 months, 2 years, and then at 5 years.

Patients are followed at 9 months, 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven node-positive breast cancer
* Postmenopausal

  * Last menstrual period more than 12 months before initial surgery OR
  * Any age with prior bilateral oophorectomy OR
  * Age 50 or over with prior hysterectomy without oophorectomy (unrelated to malignancy)
* No distant metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics

Sex:

* Female

Menopausal status:

* See Disease Characteristics

Performance status:

* WHO (ECOG) 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3 OR
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin normal
* SGOT and SGPT no greater than 1.5 times normal
* Alkaline phosphatase no greater than 1.5 times normal

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* No history of significant angina, congestive heart failure, or myocardial infarction within the past year
* No clinically significant arrhythmias or uncontrolled hypertension
* LVEF normal by MUGA, LV gated scan, or echocardiogram

Other:

* No other concurrent serious illness
* No other prior or concurrent malignancy except adequately treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-08

PRIMARY OUTCOMES:
Disease-free survival
Overall survival
Incidence of thromboembolic events during the first 9 months after randomization

SECONDARY OUTCOMES:
Tolerability
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: R. Charles Coombes, MD, MRCP, FRCP, PhD, FMedSci, Study Chair — Hammersmith Hospitals NHS Trust
Locations (1):
- Charing Cross Hospital, London, England, United Kingdom